CLINICAL TRIAL: NCT06870084
Title: The Relationship Between Masseter Muscle Thickness and Different Craniofacial Skeletal Patterns
Brief Title: Masseter Muscle Thickness and Craniofacial Skeletal Patterns
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Halil Ayyıldız, Assist. Prof., Kutahya Health Sciences University
Other Study IDs: 2023/14-28
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2023-12

CONDITIONS: Masseter; Ultrasonography; Malocclusions; Cephalometry
Keywords: masseter muscle; malocclusion; ultrasonography; cephalometry; maxillofacial development
MeSH Terms: conditions — Malocclusion | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (12):
- Class I: Patients with ANB angle between 0-4 degrees were classified as class I.
  Interventions: Other: Lateral cephalometric radiography
- Class II: Patients with ANB angle greater than 4 degrees were classified as class II.
  Interventions: Other: Lateral cephalometric radiography
- Class III: Patients with ANB angle less than 0 degrees were classified as class III.
  Interventions: Other: Lateral cephalometric radiography
- Normodivergent: Patients with SN/GoGn angle between 28 and 36 were classified as normodivergent.
  Interventions: Other: Lateral cephalometric radiography
- Hyperdivergent: Patients with SN/GoGn angle greater than 36 degrees were classified as hyperdivergent.
  Interventions: Other: Lateral cephalometric radiography
- Hypodivergent: Patients with SN/GoGn angle less than 28 degrees were classified as hypodivergent.
  Interventions: Other: Lateral cephalometric radiography
- Brachyfacial: If the facial index value was less than 84%, it was classified as brachyfacial.
  Interventions: Other: Facial photograph
- Mesofacial: A facial index value between 84% and 88% was classified as mesofacial.
  Interventions: Other: Facial photograph
- Dolichofacial: If the facial index value was greater than 88%, it was classified as dolichofacial.
  Interventions: Other: Facial photograph
- Intermolar width: The intertermolar distance was measured in millimetres. This measurement was taken from the mesiopalatinal surfaces of two maxillary first permanent molars at the level of the cervical. The measurement was taken using an electronic caliper.
  Interventions: Other: Electronic caliper
- Body Mass Index: The Body Mass Index is calculated by measuring with a standardised scale and height chart.
  Interventions: Other: Weigth and Heigth
- Masseter muscle thickness
  Interventions: Other: Ultrasonography

INTERVENTIONS:
Other: Ultrasonography — The masseter muscle thickness measurements were performed in B mode of ultrasound, midline between the zygomatic arch and mandibular plane, parallel to the mandibular plane and perpendicular to the mandibular ramus. Prior to the examination being performed in the resting position, the patient was instructed to make minimal contact between the lips without the teeth touching each other.The first USG image was recorded in this position. The patient was then requested to clench their teeth as firmly as possible, after which a second USG image was recorded from the same area. The thickness of the muscles was measured again on second recorded images. To ensure the reliability of the measurements, these procedures were repeated by the same researcher after the patients rested for five minutes.
  Groups: Masseter muscle thickness
Other: Lateral cephalometric radiography — Standard lateral cephalometric radiographs were obtained from the patients.
  Groups: Class I; Class II; Class III; Hyperdivergent; Hypodivergent; Normodivergent
Other: Facial photograph — Standard facial photographs were taken from a distance of 1.5 metres.
  Groups: Brachyfacial; Dolichofacial; Mesofacial
Other: Weigth and Heigth — The Body Mass Index is calculated by measuring with a standardised scale and height chart.
  Groups: Body Mass Index
Other: Electronic caliper — The intermaxillary distance is measured from the cervical level of the palatal surfaces of the first permanent molars to their mesial corners using an electronic caliper.
  Groups: Intermolar width

SUMMARY:
Facial morphology is influenced by hard and soft tissues, including bone and muscle. While numerous factors can lead to changes in bone tissue, soft tissues such as muscle also have an important influence. It is widely acknowledged that the function, shape and thickness of masticatory muscles have substantial effects on facial morphology and skeletal development, and are correlate with other anthropometric variables. Furthermore, a correlation has been observed between masseter muscle thickness and various characteristics of the dental arches, such as alveolar process thickness and intermaxillary width.

The evaluation of soft tissue in the region of the face is a more challenging process in comparison to that of hard tissue.The recent development of cone beam computed tomography has improved the analysis of three-dimensional skeletal morphology and jaw. However, the radiographic assessment of soft tissue remains more difficult.The thickness of masticatory muscles can be measured using computerised tomography; however, this has the disadvantage of exposing the patient to radiation. Magnetic resonance imaging (MRI) is an imaging technique that can be used to assess soft tissues. However, this technique is expensive and time-consuming. Furthermore, MRI is a static rather than a dynamic imaging technique, which makes it difficult to analyse during muscle contraction and relaxation. Ultrasound is a technique that provides dynamic imaging that can assess the masticatory muscles without the use of ionising radiation.

There are many publications in the literature that indicate that malocclusions in the vertical and sagittal dimensions can be assessed with measurements from lateral cephalometric radiographs.

ELIGIBILITY:
Inclusion Criteria: Patients who

* Patients who were 18 years of age or older,
* had skeletal malocclusion,
* were systemically healthy,
* were not taking any medication,
* had no missing teeth except for the third molars,
* had no history of congenital and/or acquired anomalies in the lips, mouth and facial regions,
* had not received orthodontic treatment before

Exclusion Criteria: Patients who

* were younger than 18 years of age
* were with systemic disease,
* used antidepressant drugs before,
* has bruxism habit,
* had orthodontic treatment or has active orthodontic treatment,
* had history of trauma and surgery in the maxillofacial region

Min Age: 18 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy patients with orthodontic malocclusion were included in the study.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
The correlation between masseter muscle thickness and sagittal skeletal malocclusions | Just at the enrollment of the patients
  The masseter muscle was measured in millimetres using ultrasound, while different skeletal malocclusions were classified using the angles between anatomical landmarks on lateral cephalometric radiographs. Intertermolar distance was measured in millimetres using an electronic caliper intraorally in the clinic. Facial index was calculated and classified using standard facial photographs, with millimetre measurements obtained using ImageJ software. The patients' height and weight were measured in centimetres and kilograms, respectively, and their body mass index was calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Science University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Togninalli D, Antonarakis GS, Papadopoulou AK. Relationship between craniofacial skeletal patterns and anatomic characteristics of masticatory muscles: a systematic review and meta-analysis. Prog Orthod. 2024 Sep 9;25(1):36. doi: 10.1186/s40510-024-00534-2. PMID 39245691